CLINICAL TRIAL: NCT06624813
Title: Partial Robot-assisted Laparoscopic Prostatectomy for Intermediate Risk Prostate Cancer
Brief Title: Partial Prostatectomy for Prostate Cancer
Acronym: P-RALP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICESP (CCEP ICESP 4017/23); BRAZILIAN MINISTRY OF HEALTH (Other: ICESP)
Record Dates: First submitted 2024-04-19; First posted 2024-10-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-03

CONDITIONS: Prostate Cancer
Keywords: partial prostatectomy in prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Partial prostatectomy (Experimental): Robot-assisted partial prostatectomy in patients with prostate cancer
  Interventions: Procedure: Robot-assisted partial prostatectomy

INTERVENTIONS:
Procedure: Robot-assisted partial prostatectomy — Focal therapy with surgery for single lobe prostate cancer, partial robot-assisted partial prostatectomy
  Other Names: Robot-assisted partial prostatectomy in patients with prostate cancer

SUMMARY:
A phase 2 study investigation of safety and feasibility of partial prostatectomy for localized prostate cancer of intermediate risk at ICESP. It will be included 50 patients that have coincident findings of prostate cancer site on prostate biopsy and a suspicious area in the magnetic resonance imaging of the prostate (PIRADS 3, 4 or 5).

DETAILED DESCRIPTION:
This Phase 2 study aims to evaluate the feasibility and standardization of robotic partial prostatectomy in patients with localized intermediate-risk prostate cancer. The study will enroll 50 patients who have undergone prostate biopsies, categorized as Gleason grade group 2 or 3, with image-guided fusion at the Cancer Institute of the State of São Paulo. Eligible patients must also have a multiparametric prostate MRI (mpMRI) with a PIRADS score of 3 to 5, consistent with the biopsy laterality.

Surgeries will be performed at the Cancer Institute of the State of São Paulo by a high-volume robotic surgeon (Rafael Ferreira Coelho) using the da Vinci surgical system. Patients involved in this research will receive follow-up care in a specialized outpatient clinic, where multidisciplinary teams will administer questionnaires assessing urinary function, sexual function, perioperative pain, and quality of life, both preoperatively and postoperatively. Data will be collected in person and stored on the online REDCap® platform.

Postoperative complications will be classified and assessed using the Clavien-Dindo scale during the first 90 days following surgery. Oncological follow-up will include quarterly PSA tests in the first year, every four months in the second year, and semi-annually from the third year onward, continuing until the end of the five-year follow-up period. A new mpMRI and protocol biopsy of the remaining prostate lobe will be performed at the 6th and 12th month of follow-up, respectively.

Patients with negative biopsies for residual neoplasia will continue to be monitored with PSA. If residual neoplasia is detected, complementary treatment will be administered based on a shared decision-making process between the physician and the patient. This study will be conducted in compliance with Resolution 466/2012 of the National Health Council/Ministry of Health (CNS/MS) and the Declaration of Helsinki (2000), following approval from the Research Ethics Committee on Human Beings (CEPSH).

The study anticipates that patients treated under this protocol will achieve satisfactory oncological outcomes, with minimal impact on functional aspects such as urinary incontinence or sexual dysfunction, and low rates of postoperative complications or negative effects on quality of life.

ELIGIBILITY:
Inclusion Criteria:

Patients with prostate cancer that presents an institutional (ICESP) fusion biopsy (cognitive or target) that presents

1. Fusion-guided prostate biopsy with mpMRI performed at the São Paulo State Cancer Institute, which
2. Present fragments for ISUP group grade (GG) ≤ 3 in only one of the prostate lobes
3. Multiparametric prostate resonance with PIRADS 3 - 5 and which is in agreement with the laterality of the tumor in the prostate biopsy
4. Life expectancy ≥ 10 years according to the Charlson score
5. Absence of second primary cancer under active treatment. Patients treated for cancer from other sites for more than 5 years and without evidence of disease will be allowed
6. Able to read, understand and complete the informed consent related to the research, as well as the research questionnaires on quality of life and functional parameters on erection and urinary continence

Exclusion Criteria:

1. Patients with prostate cancer with an histology different from adenocarcinoma
2. Suspicion of lymph node metastasis on mpMRI or distant bone scintigraphy
3. definitive signs of extraprostatic extension on mpMRI
4. history of pelvic/prostatic radiotherapy
5. ISUP grade group ≥ 4
6. Laterality of prostate biopsy discordant with mpMRI findings

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Five-year postoperative retreatment-free survival | 5 years
  Rate of patients who are free from additional treatment for the reminiscent prostatic lobe

SECONDARY OUTCOMES:
Sexual Health Inventory for Men (SHIM) | 3rd, 6th, 12th, 18th and 24th months
  - Each question is scored from 1 to 5, with the total score ranging from 5 to 25. Higher scores indicate better erectile function.
American Urological Association Symptom Index - International Prostate Symptom Score (AUA-IPSS) | 3rd, 6th, 12th, 18th and 24th months
  - Each symptom question is scored from 0 to 5, with the total symptom score ranging from 0 to 35. Higher scores indicate more Lower Urinary Tract Symptoms;
Expanded Prostate Cancer Index Composite | 3rd, 6th, 12th, 18th and 24th months
  - EPIC is a comprehensive questionnaire designed to assess the health-related quality of life in men undergoing treatment for prostate cancer. EPIC evaluates a broad range of symptoms and concerns that men may experience before, during, and after treatment. It provides a detailed assessment of urinary, bowel, sexual, and hormonal domains, each of which is scored and can be transformed to a scale of 0 to 100. Higher scores indicate better health-related quality of life or fewer symptoms.
Quality of life: EuroQol-5D | 3rd, 6th, 12th, 18th and 24th months
  EuroQol, often referred to as EQ-5D, is a standardized instrument developed by the EuroQol Group to measure health-related quality of life.
  EQ-5D: The responses to the five dimensions can be combined into a single index value representing the health status. The resulting index value reflects the health-related quality of life on a scale from less than 0 to 1, where 1 represents perfect health, 0 represents a health state equivalent to being dead, and negative values represent health states perceived as worse than being dead.
prostate specific antigen kinetics | 3rd, 6th, 12th, 18th, 24th, 30th, 36th, 42th, 48th, 54 and 60 months
  - PSA blood levels, measured by ng/mL
new magnetic resonance imaging per protocol at 6th month | 6th month
  Magnetic resonance imaging (MRI) reporting PIRADS score (Prostate Imaging-Reporting and Data System), categorical classification from 1 to 5, higher values meaning higher probability of a clinically significant prostate cancer
new postoperative prostate biopsy on the residual prostatic lobe | 12th month
  Classified as negative for neoplasia or according with the ISUP (International Society of Urological Pathology) classification system, also known as the ISUP Gleason grade group. It is a refined method for grading prostate cancer based on its microscopic appearance. It categorizes prostate cancer into five grade groups, ranging from Grade Group 1 (least aggressive, corresponding to Gleason score ≤ 6) to Grade Group 5 (most aggressive, corresponding to Gleason scores 9-10). This classification helps predict the cancer's aggressiveness and guides treatment decisions, with lower grade groups often managed with active surveillance and higher grade groups requiring more aggressive treatment due to higher risks of progression and metastasis.
Postoperative complications within 90 days of surgery | 90 days
  Number of participants with treatment-related adverse events as assessed by Calvin-Dindo classification

CONTACTS AND LOCATIONS:
Locations (1):
- Insituto do Câncer do Estado de São Paulo, São Paulo, Brazil